CLINICAL TRIAL: NCT07072325
Title: A Clinical Study Assessing the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of CD-001 in Patients With Advanced Head & Neck Cancers
Brief Title: Safety, Tolerability, PK, and Efficacy of CD-001 in Advanced Head & Neck Cancers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025(666)
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Malignant Neoplasm; Head &Amp; Neck Cancer; Head and Neck Cancer; Advanced Head and Neck Carcinoma
Keywords: head and neck cancer
MeSH Terms: conditions — Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Cohort (Experimental): CD-001 administered as an intravenous (lV) infusion
  Interventions: Drug: CD-001

INTERVENTIONS:
Drug: CD-001 — CD-001 administered as an intravenous (lV)infusion.

SUMMARY:
The goal of this prospective, single-center, open-label, dose-escalation study is to evaluate the safety, tolerability, and preliminary efficacy of CD-001 in patients with advanced head and neck cancers who have experienced disease progression (PD) or intolerance to standard systemic therapy (or lack thereof). The main question[s] it aims to answer:

* What is the safety and tolerability profile of CD-001 across escalating doses?
* What is the preliminary efficacy of CD-001 in this patient population?

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years , regardless of gender.
2. Patients with advanced head and neck cancer that are histologically or cytological confirmed, lacking standard therapy, progressing after adequate standard therapy, or intolerant of standard therapy.
3. ECOG score ≤ 2.
4. At least one measurable lesion as defined by RECIST v1.1.
5. Expected survival ≥ 3 months.

Exclusion Criteria:

1. Patients with known active central nervous system (CNS) and/or leptomeningeal metastases .
2. Patients who have undergone major organ surgery within 4 weeks prior to the first dosing, or who are expected to require major surgery during this study, or who have severe unhealed wounds, trauma, ulcers, etc.
3. Patients who have previously undergone a major organ transplant, bone marrow transplant, or allogeneic stem-cell transplant.
4. Patients who have a past or current history of active or chronic autoimmune disease and who have required systemic therapy within the past 2 years or is receiving systemic therapy for an autoimmune or inflammatory disease.
5. Patients who have received anti-tumor therapy within 4 weeks or 5 drug half-lives (whichever is shorter) prior to the first dosing.
6. At screening as determined by the investigator, the presence of any serious or uncontrollable disease or associated risk.
7. Patients with a history of ≥ Grade 3 (CTCAE) immune-related adverse events (irAEs) during prior anti-tumor therapy or permanent drug discontinuation due to irAEs.
8. Patients who have had a pulmonary embolism within 6 months prior to first dosing or have interstitial pneumonia at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | up to 12 months
  Adverse events defined as the number of participants with adverse events according

SECONDARY OUTCOMES:
Objective response rate | up to 12 months
  ORR is defined as the percentage of patients who achieve a response, which can either be complete response (complete disappearance of lesions) or partial response (reduction in the sum of maximal tumor diameters by at least 30% or more)
Progress-Free Survival | up to 12 months
  PFS is defined as the time from the administration of the first dose to first disease
Overall Survival | up to 12 months
  OS is defined as the time from the administration of the first dose to death.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cieri N, Camisa B, Cocchiarella F, Forcato M, Oliveira G, Provasi E, Bondanza A, Bordignon C, Peccatori J, Ciceri F, Lupo-Stanghellini MT, Mavilio F, Mondino A, Bicciato S, Recchia A, Bonini C. IL-7 and IL-15 instruct the generation of human memory stem T cells from naive precursors. Blood. 2013 Jan 24;121(4):573-84. doi: 10.1182/blood-2012-05-431718. Epub 2012 Nov 15. PMID 23160470
- [Background] Sabatino M, Hu J, Sommariva M, Gautam S, Fellowes V, Hocker JD, Dougherty S, Qin H, Klebanoff CA, Fry TJ, Gress RE, Kochenderfer JN, Stroncek DF, Ji Y, Gattinoni L. Generation of clinical-grade CD19-specific CAR-modified CD8+ memory stem cells for the treatment of human B-cell malignancies. Blood. 2016 Jul 28;128(4):519-28. doi: 10.1182/blood-2015-11-683847. Epub 2016 May 25. PMID 27226436
- [Background] Alvarez-Fernandez C, Escriba-Garcia L, Vidal S, Sierra J, Briones J. A short CD3/CD28 costimulation combined with IL-21 enhance the generation of human memory stem T cells for adoptive immunotherapy. J Transl Med. 2016 Jul 19;14(1):214. doi: 10.1186/s12967-016-0973-y. PMID 27435312
- [Background] Moroz A, Eppolito C, Li Q, Tao J, Clegg CH, Shrikant PA. IL-21 enhances and sustains CD8+ T cell responses to achieve durable tumor immunity: comparative evaluation of IL-2, IL-15, and IL-21. J Immunol. 2004 Jul 15;173(2):900-9. doi: 10.4049/jimmunol.173.2.900. PMID 15240677
- [Background] Hinrichs CS, Spolski R, Paulos CM, Gattinoni L, Kerstann KW, Palmer DC, Klebanoff CA, Rosenberg SA, Leonard WJ, Restifo NP. IL-2 and IL-21 confer opposing differentiation programs to CD8+ T cells for adoptive immunotherapy. Blood. 2008 Jun 1;111(11):5326-33. doi: 10.1182/blood-2007-09-113050. Epub 2008 Feb 14. PMID 18276844
- [Background] Valbon SF, Condotta SA, Richer MJ. Regulation of effector and memory CD8(+) T cell function by inflammatory cytokines. Cytokine. 2016 Jun;82:16-23. doi: 10.1016/j.cyto.2015.11.013. Epub 2015 Dec 10. PMID 26688544
- [Background] Kim TK, Herbst RS, Chen L. Defining and Understanding Adaptive Resistance in Cancer Immunotherapy. Trends Immunol. 2018 Aug;39(8):624-631. doi: 10.1016/j.it.2018.05.001. Epub 2018 May 22. PMID 29802087
- [Background] Zappasodi R, Merghoub T, Wolchok JD. Emerging Concepts for Immune Checkpoint Blockade-Based Combination Therapies. Cancer Cell. 2018 Apr 9;33(4):581-598. doi: 10.1016/j.ccell.2018.03.005. PMID 29634946
- [Background] Jenkins RW, Barbie DA, Flaherty KT. Mechanisms of resistance to immune checkpoint inhibitors. Br J Cancer. 2018 Jan;118(1):9-16. doi: 10.1038/bjc.2017.434. Epub 2018 Jan 2. PMID 29319049
- [Background] Helmink BA, Gaudreau PO, Wargo JA. Immune Checkpoint Blockade across the Cancer Care Continuum. Immunity. 2018 Jun 19;48(6):1077-1080. doi: 10.1016/j.immuni.2018.06.003. PMID 29924973
- [Background] Huang AC, Postow MA, Orlowski RJ, Mick R, Bengsch B, Manne S, Xu W, Harmon S, Giles JR, Wenz B, Adamow M, Kuk D, Panageas KS, Carrera C, Wong P, Quagliarello F, Wubbenhorst B, D'Andrea K, Pauken KE, Herati RS, Staupe RP, Schenkel JM, McGettigan S, Kothari S, George SM, Vonderheide RH, Amaravadi RK, Karakousis GC, Schuchter LM, Xu X, Nathanson KL, Wolchok JD, Gangadhar TC, Wherry EJ. T-cell invigoration to tumour burden ratio associated with anti-PD-1 response. Nature. 2017 May 4;545(7652):60-65. doi: 10.1038/nature22079. Epub 2017 Apr 10. PMID 28397821
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751